CLINICAL TRIAL: NCT02242708
Title: The Effectiveness of Autonomic Nervous System, Sleep Quality, and Immune Regulation for Shift Nurses Practicing Alternative Nostril Breathing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Bing Show Chwan Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ming-Ho Lee, MD., Chang Bing Show Chwan Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1010807
Record Dates: First submitted 2014-09-15; First posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Shift Nurses

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal breathing (No Intervention): The control group will do normal breathing.
- Alternative nostril breathing (Experimental): The experimental groups will do alternative nostril breathing twice a week (20 minutes/time) for 3 months.
  Interventions: Behavioral: Alternative nostril breathing

INTERVENTIONS:
Behavioral: Alternative nostril breathing — The experimental groups will do alternative nostril breathing twice a week (20 minutes/time) for 3 months.
  Arms: Alternative nostril breathing

SUMMARY:
The purpose of this study is to evaluate the efficacy of shift nurses practicing alternative nostril breathing to improve life quality, autonomic nervous system and immune status.

DETAILED DESCRIPTION:
Breathing is regulated by autonomic nervous system. It is well-known that breathing exercise can regulate autonomic nervous function and promote relaxation. However, the mechanism for better immunity and sleep quality is not clear. We postulate that alternative nostril breathing might benefit nurses after undergoing shift work. The benefits could be due to improvement of autonomic nervous function, sleep quality, and even immune function.

The study design will include a randomization of two groups, with a control group and one experimental groups for 3 months (12 weeks). The control group will do normal breathing. The experimental groups will do alternative nostril breathing twice a week (20 minutes/time) for 3 months.

The study primary endpoints are 1) to improve autonomic nervous function, 2) to improve sleep quality and 3) to enhance human immunity.

We anticipate to reach the primary endpoints and publish the primary results in one year.

ELIGIBILITY:
Inclusion Criteria:

* Shift nurses

Exclusion Criteria:

* Upper respiratory tract infection such as nasal congestion, runny nose, coughing, wheezing, nosebleeds, fever and other symptoms.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Improve sleep quality. | Change from baseline in sleep quality at 3 months.
  Sleep quality will be assessed by pittsburg sleep quality index at three different times: (1)baseline data: before alternate nostril breathing practice ,(2)outcome data:6 and 12 weeks alternate nostril breathing practice, right after exercise measures post-test.

SECONDARY OUTCOMES:
Enhance human immunity | Change from baseline in human immunity at 3 months.
  Lymphocytes will be extracted from peripheral blood for analyses of lymphocytes subpopulation, polarization and its related cytokines. Saliva will be collected at 3 different times: (1)baseline data: before alternate nostril breathing program ,(2)outcome data:6 and 12 weeks alternate nostril breathing practice, right after exercise measures post-test.
Improve autonomic nervous function | Change from baseline in autonomic nervous function at 3 months.
  Autonomic nervous function will be assessed by biofeedback index using heart rate variability at three different times: (1)baseline data: before alternate nostril breathing practice ,(2)outcome data:6 and 12 weeks alternate nostril breathing practice, right after exercise measures post-test.

CONTACTS AND LOCATIONS:
Overall Officials: Kuender D. Yang, PhD, Study Director — Chang Bing Show Chwan Memorial Hospital; Ming-Ho Lee, Principal Investigator — Chang Bing Show Chwan Memorial Hospital
Locations (1):
- Division of Core Laboratory; Chang Bing Show Chwan Memorial Hospital, Changhua County, Taiwan